CLINICAL TRIAL: NCT06795399
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Proof of Concept Trial for OPC-131461 in Patients Hospitalized for Worsening Heart Failure With Laboratory Evidence of Incomplete Decongestion Following Urgent Decongestive Therapy
Brief Title: A Proof-of-concept Trial for OPC 131461 in Patients Hospitalized for Worsening Heart Failure
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 351-201-00015
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- OPC-131461 5 mg (Experimental): Participants will receive OPC-131461 5 mg, orally, once daily for 30 days.
  Interventions: Drug: OPC-131461
- OPC-131461 10 mg (Experimental): Participants will receive OPC-131461 10 mg, orally, once daily for 30 days.
  Interventions: Drug: OPC-131461
- Placebo (Placebo Comparator): Participants will receive OPC-131461 matched placebo, orally, once daily for 30 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OPC-131461 — OPC-131461 will be administered as oral tablets.
  Arms: OPC-131461 10 mg; OPC-131461 5 mg
Drug: Placebo — OPC-131461 matched placebo will be administered as oral tablets.
  Arms: Placebo

SUMMARY:
The primary objective of the study is to compare relative changes in blood N-terminal pro-B-type natriuretic peptide (NT-proBNP) levels after 30 days of treatment in participants with worsening heart failure (WHF), who are treated with either OPC-131461 or placebo.

DETAILED DESCRIPTION:
Each participant in this trial is expected to participate in the following periods of the trial:

* Screening/qualification period: up to 48 hours (2 days)
* Double-blind treatment period: 30 days
* Safety follow-up period: 7 days
* Vital status follow-up period: 6 months

Eligible participants will be randomized to receive the study drug (1 of 2 dose levels [5 milligrams (mg) or 10 mg] of OPC-131461 tablets or placebo) in a 1:1:1 ratio.

Overall, the trial duration is expected to be approximately 210 days (7 months).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HF ≥ 3 months prior to screening.
* Admitted to the hospital with primary diagnosis of WHF and received treatment with intravenous (IV) diuretics.
* Eligible participants will be randomized no earlier than 48 hours and up to 5 days after presentation to the hospital as long as they meet the following definition of stable status: Stable for at least 24 hours, defined by systolic blood pressure (SBP) ≥ 90 millimeters of mercury (mmHg) for preceding 24 hours, no increase in diuretic dose for 24 hours prior to randomization, did not receive IV inotropic or vasodilator (including nitrates) for 24 hours prior to randomization, and no oxygen therapy or mechanical ventilation in the 24 hours prior to randomization
* Left ventricular ejection fraction (LVEF) assessed either during hospitalization for Index Event or within 12 months prior to randomization.
* Has evidence of incomplete decongestion, indicated by NT-proBNP levels > 750 picograms per milliliter (pg/mL) (or > 1000 pg/mL if in atrial fibrillation). At hospital sites where NT proBNP test is unavailable at screening: B-type natriuretic peptide (BNP) > 375 pg/mL (or > 500 pg/mL if in atrial fibrillation).

Exclusion Criteria:

* Primary cause of WHF (Index Event) due to valvular heart disease (defined as severe aortic or primary mitral regurgitation, moderate or severe aortic stenosis, any mitral stenosis requiring surgical repair, or active endocarditis), congenital heart disease, hypertrophic obstructive cardiomyopathy, pulmonary embolism, Type I myocardial infarction, infection, severe anemia, exacerbation of chronic obstructive pulmonary disease (COPD), or sustained ventricular tachycardia, or bradycardia with sustained ventricular rate < 45 beats/minute.
* Duration of hospitalization for Index Event > 2 weeks at time of screening.
* End-stage HF requiring at the time of screening left ventricular assist device (LVAD), intra-aortic balloon pump (IABP) or any similar mechanical support.
* Cardiac surgery (coronary artery bypass grafting [CABG]), percutaneous coronary intervention (PCI), implantation of a cardiac device or cardiac mechanical support implantation within 30 days prior to randomization or planned during the study
* Severely impaired renal function eGFR < 25 milliliters per minute per 1.73-meter square (mL/min/1.73m^2).
* History of dialysis or kidney transplant.
* History of cirrhosis or noncirrhotic portal hypertension.
* Severe hyponatremia Sodium (Na) level < 125 mEq/L (milliequivalents per liter) or hypernatremia Na level > 145 mEq/L).
* Systolic blood pressure < 90 mmHg at screening.
* History of or current hepatitis or acquired immunodeficiency syndrome or carriers of hepatitis B surface antigen (HBsAg) and/or hepatitis C antibodies (anti-HCV), or human immunodeficiency virus (HIV) antibodies.
* History of any significant drug allergy or known or suspected hypersensitivity to any component of the study drug.
* Use of any investigational drug within 30 days prior to screening.
* History of serious mental disorders that, in the opinion of the investigator, would exclude the participant from participating in this trial.

Note: Other protocol-specified inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Proportional Change From Baseline in Serum Concentration of NT-proBNP at Day 31 | Baseline, Day 31
  Proportional change from baseline in serum concentration of NT-proBNP is defined as the ratio of NT-proBNP at Day 31 over baseline.

SECONDARY OUTCOMES:
Proportional Change From Baseline in Serum Concentration of NT-proBNP at Days 8 and 15 | Baseline, Days 8 and 15
  Proportional change from baseline in serum concentration of NT-proBNP is defined as the ratio of NT-proBNP at Day 8 over baseline and at Day 15 over baseline.
Time to First Heart Failure (HF) Rehospitalization | From first dose of study drug up to end of treatment period (up to 30 days)
Time to First Urgent HF Outpatient Visit | From first dose of study drug up to end of treatment period (up to 30 days)
Time to Cardiovascular (CV) Death | From first dose of study drug up to end of treatment period (up to 30 days)
Composite Endpoint Defined by the Win Ratio | From the first dose of the study drug up to end of treatment period (up to 30 days)
  A hierarchical composite of CV death, number of HF rehospitalizations, number of urgent HF outpatient visits, time to first HF rehospitalization or urgent HF outpatient visit, and change from baseline in Kansas City Cardiomyopathy Questionnaire - 23 items (KCCQ-23) Total Symptom Score (difference larger or equal to 5) will be analyzed using the Win ratio method.
Change From Baseline in Kansas City Cardiomyopathy Questionnaire - 23 items (KCCQ-23) Clinical Summary Score | Up to 31 days
  The KCCQ-23 is a questionnaire consisting of 23 items to measure health status, symptoms, and quality of life in participants with heart failure. The KCCQ-23 consists of the following domains: Physical Limitation, Symptoms, Self-efficacy and knowledge, Quality of Life, Social Limitation. A functional status score is calculated from physical limitations and symptoms. The clinical summary score is derived from the functional status score, quality of life, and social limitations domains and range from 0-100. A higher score indicates fewer symptoms and better physical functioning, reflecting improved overall clinical status.
Change From Baseline in KCCQ-23 Total Symptom Score | Up to 31 days
  The KCCQ-23 is a questionnaire consisting of 23 items to measure health status, symptoms, and quality of life in participants with heart failure. The KCCQ-23 consists of the following domains: Physical Limitation, Symptoms, Self-efficacy and knowledge, Quality of Life, Social Limitation. The total symptom score combines responses from the symptom frequency and symptom burden domains. Score ranges from 0-100, where higher scores indicate fewer symptoms and a better symptom experience.
Change From Baseline in KCCQ-23 Physical Limitations Score | Up to 31 days
  The KCCQ-23 is a questionnaire consisting of 23 items to measure health status, symptoms, and quality of life in participants with heart failure. The KCCQ-23 consists of the following domains: Physical Limitation, Symptoms, Self-efficacy and knowledge, Quality of Life, Social Limitation. The Physical Limitation Score will assess the impact of HF on participants' ability to perform physical activities. Scores range from 0-100, with higher scores reflecting fewer physical limitations and better functional capacity.
Change From Baseline in Body Weight | Up to 37 days
Change From Baseline in EVEREST Congestion Score | Up to 37 days
  The EVEREST Congestion Score will assess the severity of congestion in participants with HF. The score includes clinical signs and symptoms such as edema, dyspnea, orthopnea, jugular vein distention, rales, and fatigue. The total score ranges from 0-18, with a higher score indicating greater severity of congestion and a lower score reflecting less congestion and improvement in symptoms.
Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) | Up to 37 days
Number of Participants With Serum Electrolyte Abnormalities | Up to 37 days
Number of Participants With Hypotension/Orthostatic Hypotension and Related Treatment-emergent Adverse Events (TEAEs) of Syncope and Presyncope | Up to 37 days
Number of Participants With Major and Minor Bleeding Events | Up to 37 days

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com
URL: http://clinical-trials.otsuka.com